CLINICAL TRIAL: NCT03078075
Title: NIDA (National Institute on Drug Abuse) CTN (Clinical Trials Network) Protocol 0068: Accelerated Development of Additive Pharmacotherapy Treatment (ADAPT-2) for Methamphetamine Use Disorder
Brief Title: Accelerated Development of Additive Pharmacotherapy Treatment (ADAPT-2) for Methamphetamine Use Disorder
Acronym: ADAPT-2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); The Emmes Company, LLC (Industry)
Responsible Party: Principal Investigator, Madhukar H. Trivedi, MD, Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CTN-0068; UG1DA020024 (NIH)
Record Dates: First submitted 2017-03-02; First posted 2017-03-13 (Actual); Results first posted 2021-03-29 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Methamphetamine Use Disorder
Keywords: Methamphetamine; Methamphetamine Use Disorder; Naltrexone; Bupropion; Vivitrol®
MeSH Terms: interventions — phospholamban; Injections

STUDY DESIGN:
Intervention Model Description: During the study, participants may or may not be switched to another group due to the adaptive aspect of the study design. Participants appearing to respond well to their original treatment assignment will not be switched.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active Medication Combination (AMC) (Experimental): injectable extended release naltrexone plus once daily oral extended-release bupropion tablets
  Interventions: Drug: Naltrexone: Vivitrol®; Drug: Bupropion: Wellbutrin XL®
- Matched Placebo (PLB) (Placebo Comparator): injectable matching placebo plus once-daily oral placebo tablets
  Interventions: Drug: Placebo (PLB) Injectable; Drug: Placebo (PLB) Oral

INTERVENTIONS:
Drug: Naltrexone: Vivitrol® — Naltrexone: 380 mg vial, 4 intramuscular injections administered every 3 weeks
  Other Names: Arm: Experimental - Active Medication Combination (AMC)
  Arms: Active Medication Combination (AMC)
Drug: Placebo (PLB) Injectable — Placebo: 4 intramuscular injections administered every 3 weeks
  Other Names: Injectable matching (to Naltrexone) placebo; Arm: Placebo Comparator - matched Placebo (PLB)
  Arms: Matched Placebo (PLB)
Drug: Bupropion: Wellbutrin XL® — Bupropion: 450 mg oral dose daily
  Other Names: Arm: Experimental - Active Medication Combination (AMC)
  Arms: Active Medication Combination (AMC)
Drug: Placebo (PLB) Oral — Placebo: once-daily oral placebo tablets
  Other Names: Oral matching (to Bupropion) placebo tablets; Arm: Placebo Comparator - matched Placebo (PLB)
  Arms: Matched Placebo (PLB)

SUMMARY:
This is a double-blind, placebo-controlled, randomized clinical trial evaluating the efficacy of extended-release naltrexone plus bupropion as a combination pharmacotherapy for methamphetamine use disorder. Participants will be randomly assigned to the active medication combination (AMC) group or matching placebo group and will receive medications over the course of 12 weeks. Follow-ups will occur in weeks 13 and 16.

DETAILED DESCRIPTION:
There will be 400 adults with moderate or severe methamphetamine use disorder randomized into this multi-site study. Eligibility will be determined during a maximum 21 day screening period. After screening is completed and eligibility is confirmed, including successful administration of a naloxone challenge, participants will begin the 12 week medication phase of the trial. Participants will be randomized to either the 1) AMC arm and receive injections of extended release naltrexone (XR-NTX; as Vivitrol®) plus once-daily oral extended-release bupropion tablets (BUP-XL) or the 2) matching placebo (PLB) arm and receive injections of placebo (iPLB) plus once-daily oral placebo (oPLB) tablets. During the course of the study, participants may be switched to another arm, as determined by the a priori adaptive aspect of the study design. Participants appearing to respond well to their original treatment assignment will not be switched. Overall, approximately 50% of the participants will receive the AMC. Injections will be administered every three weeks, in weeks 1, 4, 7, and 10. Take-home oral study medication (BUP-XL or oPLB) will be dispensed weekly for dosing on non-clinic days. Participants will be asked to attend the clinic twice weekly for observed oral medication dosing, assessments, collection of urine samples, and once-weekly medical management. On non-clinic days, participants will participate in smartphone app-based medication adherence activities. Participants will be asked to complete assessments as indicated on the schedule of assessments. Following the 12 week medication phase, participants will complete a follow-up phase, including a medication taper and post-medication phase follow-up visits during weeks 13 and 16.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 65 years old;
* Interested in reducing/stopping methamphetamine use;
* Speak English;
* Agree to use acceptable birth control (if applicable);
* Be opioid-free at randomization;
* Willing to comply with all study procedures and medication instructions;
* Agree to use a cell phone (or similar study device) to take videos of medication dosing.

Exclusion Criteria:

* Medical or psychiatric condition which would make participation unsafe;
* Recently participated in a study of pharmacological or behavioral treatment for methamphetamine use disorder;
* Recently taken an investigational drug;
* Prescribed and taken naltrexone or bupropion ≤ 30 days from consent;
* Current or planned extended absence during study period (e.g., jail, surgery, pending legal action);
* Currently pregnant or breastfeeding.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 403 (Actual)
Dates: Start 2017-05-05 (Actual); Primary Completion 2019-07-03 (Actual); Study Completion 2019-07-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Madhukar Trivedi, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (8):
- United States (8):
  - University of California Los Angeles (UCLA) Center for Behavioral Addiction Medicine (CBAM), Los Angeles, California
  - Substance Use Research Unit (SURU) at the San Francisco Dept. of Public Health, San Francisco, California
  - Hennepin County Medical Center- Berman Center for Research, Minneapolis, Minnesota
  - New York State Psychiatric Institute (NYSPI)- Substance Use Research Center (SURC), New York, New York
  - CODA, Inc., Portland, Oregon
  - Behavioral Health Services (BHS) of Pickens County, Pickens, South Carolina
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - University of Texas Health Science Center - Center for Neurobehavioral Research on Addiction (CNRA), Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
Data from this study will be available to researchers on the website https://datashare.nida.nih.gov/ after the study is complete and the data is analyzed. This website will not include information that can identify individual study participants.The following information will be posted: Study protocol, reference to study publication of primary outcome, data sets (SAS and ASCII ), annotated case report forms, define file (also known as Data Dictionary), study-specific de-identification notes. Prior to downloading any study data, the user will be prompted to complete a registration agreement for data use. Users will have to register a name and valid e-mail address in order to download data and to accept their responsibility for using data in accordance with the NIDA Data Share Agreement.

REFERENCES:
- [Derived] Jha MK, Ghitza UE, Shoptaw S, Minhajuddin A, Kuruvila S, Wakhlu S, Nunes EV, Schmitz J, Coffin PO, Bart G, Carmody T, Trivedi MH. Early Change in Depressive Symptom Severity With Naltrexone-Bupropion Combination and Its Association With Reduction in Methamphetamine Use in ADAPT-2 Trial. J Clin Psychiatry. 2025 Jul 30;86(3):25m15825. doi: 10.4088/JCP.25m15825. PMID 40767786
- [Derived] Li MJ, Chau B, Belin T, Carmody T, Jha MK, Marino EN, Trivedi M, Shoptaw SJ. Extended observation of reduced methamphetamine use with combined naltrexone plus bupropion in the ADAPT-2 trial. Addiction. 2024 Oct;119(10):1840-1845. doi: 10.1111/add.16529. Epub 2024 Jun 10. PMID 38856086
- [Derived] Okafor CN, Carmody T, Stotts AL, Bart G, Mayes TL, Karns-Wright T, Trivedi M, Shoptaw S, Potter JS. Sociodemographic and patient reported outcomes by racial and ethnicity status among participants in a randomized controlled trial for methamphetamine use disorder. Drug Alcohol Depend Rep. 2024 Apr 6;11:100230. doi: 10.1016/j.dadr.2024.100230. eCollection 2024 Jun. PMID 38665252
- [Derived] Trombello JM, Kulikova A, Mayes TL, Nandy K, Carmody T, Bart G, Nunes EV, Schmitz J, Kalmin M, Shoptaw S, Trivedi MH. Psychometrics of the Concise Health Risk Tracking Self-Report (CHRT-SR16) Assessment of Suicidality in a Sample of Adults with Moderate to Severe Methamphetamine Use Disorder: Findings from the ADAPT-2 Randomized Trial. Neuropsychiatr Dis Treat. 2023 Jun 22;19:1443-1454. doi: 10.2147/NDT.S406909. eCollection 2023. PMID 37377462
- [Derived] Vo HT, Kulikova A, Mayes TL, Carmody T, Shoptaw S, Ling W, Trombello JM, Trivedi MH. Psychometric properties of the Treatment Effectiveness Assessment in methamphetamine use disorder. J Subst Use Addict Treat. 2023 Aug;151:209085. doi: 10.1016/j.josat.2023.209085. Epub 2023 May 26. PMID 37245855
- [Derived] Trivedi MH, Walker R, Ling W, Dela Cruz A, Sharma G, Carmody T, Ghitza UE, Wahle A, Kim M, Shores-Wilson K, Sparenborg S, Coffin P, Schmitz J, Wiest K, Bart G, Sonne SC, Wakhlu S, Rush AJ, Nunes EV, Shoptaw S. Bupropion and Naltrexone in Methamphetamine Use Disorder. N Engl J Med. 2021 Jan 14;384(2):140-153. doi: 10.1056/NEJMoa2020214. PMID 33497547

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All participants were randomized to either the AMC arm or the Placebo arm in Week 1; thus all are represented in the two Stage 1 categories (total 403).
  All participants also are represented in Stage 2. Some participants were re-randomized at Week 7 and some were not; thus the four Stage 2 categories also total 403.
Groups:
- Stage 1 Placebo Non-responders Re-randomized to Placebo at Stage 2: Those participants randomized to the Placebo arm in Stage 1 (Week 1) who were non-responders at week 5 and 6, and then re-randomized to Placebo at stage 2.
- Stage 1 Placebo Non-responders Re-randomized to AMC at Stage 2: Those participants randomized to the Placebo arm in Stage 1 (Week 1) who were non-responders at week 5 and 6, and then re-randomized to AMC at stage 2.
- Stage 1 Placebo Non-responders Not Re-randomized at Stage 2: Those participants randomized to the Placebo arm in Stage 1 (Week 1) who were non-responders at week 5 and 6 and then not re-randomized at stage 2, remained in the Placebo arm.
- Stage 1 Placebo Responders Not Re-randomized at Stage 2: Those participants randomized to the Placebo arm in Stage 1 (Week 1) who were responders at week 5 and 6 and then not re-randomized at stage 2, remained in the Placebo arm.
- Stage 1 AMC Remaining on AMC at Stage 2: All participants who were randomized to the Active Medication Combination arm in Stage 1 (Week 1) remained in the AMC arm throughout the study (Weeks 1-12).
Period: Overall Study
Arm/Group | Stage 1 Placebo Non-responders Re-randomized to Placebo at Stage 2 | Stage 1 Placebo Non-responders Re-randomized to AMC at Stage 2 | Stage 1 Placebo Non-responders Not Re-randomized at Stage 2 | Stage 1 Placebo Responders Not Re-randomized at Stage 2 | Stage 1 AMC Remaining on AMC at Stage 2
Started | 111 | 114 | 59 | 10 | 109
Completed | 106 | 103 | 19 | 9 | 78
Not Completed | 5 | 11 | 40 | 1 | 31

BASELINE CHARACTERISTICS:
Population: The Baseline characteristics are based on stage 1 assignment
Groups:
- Active Medication Combination (AMC): injectable extended release naltrexone plus once daily oral extended-release bupropion tablets
  Naltrexone: Vivitrol®: Naltrexone: 380 mg vial, 4 intramuscular injections administered every 3 weeks
  Bupropion: Wellbutrin XL® (Extended release): Bupropion: 450 mg oral dose daily
- Total: Total of all reporting groups
Arm/Group | Active Medication Combination (AMC) | Matched Placebo (PLB) | Total
Number analyzed (Participants) | 109 | 294 | 403
Age, Continuous [Mean (Standard Deviation); unit: years] | 41 (10.6) | 41 (10.0) | 41 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 95 | 126
  Male | 78 | 199 | 277
Race/Ethnicity, Customized [Number; unit: participants]
  Not Hispanic/ Latino | 96 | 249 | 345
  Hispanic/Latino | 13 | 42 | 55
  Unknown Ethnicity | 0 | 2 | 2
  Refused to answer Ethnicity | 0 | 1 | 1
  American Indian/Alaska Native | 2 | 4 | 6
  Asian | 1 | 10 | 11
  Black/ African American | 10 | 38 | 48
  Native Hawaiian/ Pacific Islander | 1 | 1 | 2
  White | 82 | 205 | 287
  Other Race | 6 | 14 | 20
  Multiracial | 3 | 13 | 16
  Unknown Race | 2 | 8 | 10
  Refused to answer Race | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Response During Medication Phase at Stage 1
Description: Treatment response is defined as 'Responder' and 'Non-Responder'.
  Responder : Participant who meet responder criterion by providing at least 3 out of a possible 4 methamphetamine-negative urine tests at the end of stage 1 (weeks 5-6).
  Non-Responder: All other participants without 3 or 4 methamphetamine-negative UDS (Urine Drug Screen).
Time Frame: At weeks 6
Population: Intention to treat analysis was done including drop-out
Measure: Count of Participants; unit: Participants
Groups:
- Stage 1 Placebo: Those participants randomized to the Placebo arm in Stage 1 (Week 1); these participants may or may not be re-randomized in Week 7.
- Stage 1 AMC: Those participants who were randomized to the Active Medication Combination arm in Stage 1 (Study Week 1) remained in the AMC arm throughout the study (Weeks 1-12).
Arm/Group | Stage 1 Placebo | Stage 1 AMC
Number analyzed (Participants) | 294 | 109
Participants
  Responders (Methamphetamine negative UDS results) | 10 | 18
  Non-responders (Methamphetamine positive UDS results) | 284 | 91

2. Primary Outcome: Number of Participants With Treatment Response During Medication Phase at Stage 2
Description: Treatment response is defined as 'Responder' and 'Non-Responder'.
  Responder : Participant who meet responder criterion by providing at least 3 out of a possible 4 methamphetamine-negative urine tests at the end of stage 1 (weeks 5-6).
  Non-Responder: All other participants without 3 or 4 methamphetamine-negative UDS.
Time Frame: At week 12
Measure: Count of Participants; unit: Participants
Groups:
- Stage 2 Re-Randomized Placebo: Those participants who were randomized to the Placebo arm in Stage 1 (Week 1) and were deemed Non-Responders at Study Weeks 5-6 and were re-randomized to the Placebo arm in Stage 2 (Week 7).
- Stage 2 Re-Randomized AMC: Those participants who were randomized to the Placebo arm in Stage 1 (Week 1) and were deemed Non-Responders at Study Weeks 5-6 and were re-randomized to the Active Medication Combination arm in Stage 2 (Week 7)
- Stage 2 Not Re-Randomized Placebo: Those participants who were originally randomized to the Placebo arm in Stage 1 (and may or may not have been deemed Non-Responders at Study Weeks 5-6) and were not Re-Randomized, so they remained in the Placebo arm throughout the study (Weeks 1-12).
- Stage 2 Not Re-Randomized AMC: All participants who were randomized to the Active Medication Combination arm in Stage 1 (Week 1) remained in the AMC arm throughout the study (Weeks 1-12).
Arm/Group | Stage 2 Re-Randomized Placebo | Stage 2 Re-Randomized AMC | Stage 2 Not Re-Randomized Placebo | Stage 2 Not Re-Randomized AMC
Number analyzed (Participants) | 111 | 114 | 69 | 109
Participants
  Responders (Methamphetamine negative UDS results) | 2 | 13 | 9 | 21
  Non-Responders (Methamphetamine positive UDS results) | 109 | 101 | 60 | 88

3. Secondary Outcome: Treatment Effectiveness Score of Participants at Stage 1
Description: The Treatment Effectiveness Score (TES) as measured by UDS results, during the treatment period. The TES is the percentage of the expected urine drug screens that were negative for each drug. Twelve urine drug screens are expected within each stage.
Time Frame: At weeks 6
Population: Intention to treat analysis was done including drop-out
Measure: Mean (Standard Deviation); unit: percentage of urine drug screens
Arm/Group | Stage 1 Placebo | Stage 1 AMC
Number analyzed (Participants) | 294 | 109
percentage of urine drug screens | 5.72 (13.41) | 13.84 (22.97)

4. Secondary Outcome: Treatment Effectiveness Score of Participants at Stage 2
Description: The Treatment Effectiveness Score (TES) as measured by UDS results, during the treatment period. The TES is the percentage of the expected urine drug screens that were negative for each drug. Twelve urine drug screens are expected within each stage. The range of possible scores are 0-100 and higher score indicates better outcomes.
Time Frame: At week 12
Population: As per study protocol, stage 2 secondary outcomes are reported for only re-randomized groups (Placebo and AMC)
Measure: Mean (Standard Deviation); unit: percentage of urine drug screens
Arm/Group | Stage 2 Re-Randomized Placebo | Stage 2 Re-Randomized AMC
Number analyzed (Participants) | 111 | 114
percentage of urine drug screens | 7.45 (16.02) | 11.55 (24.55)

5. Secondary Outcome: Percentage of Participants Who Used Methamphetamine in the Pre-evaluation Period
Description: Methamphetamine use, as measured by UDS (urine drug screen) in the pre-evaluation period (Weeks 1-4 for Stage 1 and Weeks 7-10 for Stage 2 )
Time Frame: Weeks 1-4 and Weeks 7-10
Population: Intention to treat analysis was done including drop-out.
Measure: Number; unit: percentage of participants
Arm/Group | Stage 1 Placebo | Stage 1 AMC | Stage 2 Re-Randomized Placebo | Stage 2 Re-Randomized AMC | Stage 2 Not Re-Randomized Placebo | Stage 2 Not Re-Randomized AMC
Number analyzed (Participants) | 294 | 109 | 111 | 114 | 69 | 109
percentage of participants | 5.10 | 11.93 | 7.95 | 10.20 | 29.46 | 22.56

6. Secondary Outcome: Mean Maximum Number of Consecutive Visits Negative UDS at Stage 1
Description: Measured by maximum consecutive negative UDS: Count the number and range 0-12 and report the maximum number.
Time Frame: At week 6
Measure: Mean (Standard Deviation); unit: UDS test results
Groups:
- Placebo: Those participants randomized to the Placebo arm in Stage 1
- AMC (Active Medication Combination Arm): Those participants who were randomized to the Active Medication Combination arm in Stage 1
Arm/Group | Placebo | AMC (Active Medication Combination Arm)
Number analyzed (Participants) | 294 | 109
UDS test results | 0.54 (1.31) | 1.37 (2.50)

7. Secondary Outcome: Mean Maximum Number of Consecutive Visits Negative UDS at Stage 2
Description: Measured by maximum consecutive negative UDS: Count the number and range 0-12 and report the maximum number.
Time Frame: Stage 2 evaluation period at Weeks 12
Measure: Mean (Standard Deviation); unit: UDS test results
Groups:
- Stage 2 Re-Randomized Placebo: Those participants randomized to the Placebo arm in Stage 2
- Stage 2 Re-Randomized AMC (Active Medication Combination Arm): Those participants who were randomized to the Active Medication Combination arm in Stage 2
Arm/Group | Stage 2 Re-Randomized Placebo | Stage 2 Re-Randomized AMC (Active Medication Combination Arm) | Stage 2 Not Re-Randomized Placebo | Stage 2 Not Re-Randomized AMC
Number analyzed (Participants) | 111 | 114 | 69 | 109
UDS test results | 0.61 (1.46) | 1.18 (2.72) | 3.10 (4.39) | 2.63 (4.13)

8. Secondary Outcome: Mean Number of Study Weeks With Two Methamphetamine-negative UDS at Stage 1
Description: Measured by the number of study weeks during the treatment period with two methamphetamine-negative UDS.
Time Frame: At week 6
Measure: Mean (Standard Deviation); unit: weeks
Groups:
- AMC (Active Medication Combination): Those participants who were randomized to the Active Medication Combination arm in Stage 1
Arm/Group | Placebo | AMC (Active Medication Combination)
Number analyzed (Participants) | 294 | 109
weeks | 0.15 (0.55) | 0.56 (1.20)

9. Secondary Outcome: Mean Number of Study Weeks With Two Methamphetamine-negative UDS at Stage 2
Description: Measured by the number of study weeks during the treatment period with two methamphetamine-negative UDS.
Time Frame: At week12
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | Stage 2 Re-Randomized Placebo | Stage 2 Re-Randomized AMC | Stage 2 Not Re-Randomized Placebo | Stage 2 Not Re-Randomized AMC
Number analyzed (Participants) | 111 | 114 | 69 | 109
weeks | 0.20 (0.70) | 0.50 (1.35) | 1.48 (2.21) | 1.20 (2.08)

10. Secondary Outcome: Mean Change of Percentage of Methamphetamine Abstinent Days Measured by Self-report at Stage 1
Description: Methamphetamine use selfreported on TLFB ( Timeline Followback) during the follow-up period.
  The baseline measure is the percentage of abstinent days in the 30 days prior to randomization. The outcome is the change in percentage of abstinent days.
Time Frame: Baseline, week 6
Measure: Mean (Standard Error); unit: percentage of abstinent days
Arm/Group | Stage 1 Placebo | Stage 1 AMC
Number analyzed (Participants) | 294 | 109
percentage of abstinent days | 14.0 (1.3) | 27.2 (2.88)

11. Secondary Outcome: Mean Change Percentage of Methamphetamine Abstinent Days Measured by Self-report at Stage 2
Description: as for outcome 10
Time Frame: week 7, week 12
Population: These numbers come from a model which does not use the Stage 2 Not rerandomized data. As per study protocol, stage 2 secondary outcomes are reported for only re-randomized groups (Placebo and AMC). Data for Not Re-Randomized groups at stage 2 were not included for the main analysis, thus not reported
Measure: Mean (Standard Error); unit: percentage of abstinent days
Arm/Group | Stage 2 Re-Randomized Placebo | Stage 2 Re-Randomized AMC
Number analyzed (Participants) | 111 | 114
percentage of abstinent days | 16 (1.5) | 25.3 (2.6)

12. Secondary Outcome: Mean Change of Methamphetamine Craving at Stage 1
Description: Severity of methamphetamine craving, as measured by Visual Analog Craving Scales (VAS), during the treatment period. VAS scores range from 0 (no craving) to 100 (most intense craving possible). The VAS is completed at screening, once a week during the treatment period, and at the follow-up visits.
Time Frame: Baseline, week 6
Population: Intention to treat analysis was done including drop-out
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Stage 1 Placebo | Stage 1 AMC
Number analyzed (Participants) | 294 | 109
score on a scale | -22.33 (1.82) | -29.98 (3.17)

13. Secondary Outcome: Mean Change of Methamphetamine Craving at Stage 2
Description: as for outcome 12
Time Frame: week 7, week 12
Population: As per study protocol, stage 2 secondary outcomes are reported for only re-randomized groups (Placebo and AMC). Data for Not Re-Randomized groups at stage 2 were not included for the main analysis, thus not reported
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Stage 2 Re-Randomized Placebo | Stage 2 Re-Randomized AMC
Number analyzed (Participants) | 111 | 114
score on a scale | -20.52 (1.72) | -31.79 (3.17)

14. Secondary Outcome: Mean Number of Abstinent Days of Participants Who Used Other Substance Measured by UDS at Stage 1
Description: Other substance use including Amphetamine, Non-Methamphetamine Drug, Cocaine, Alcohol, Cigarettes, as measured by UDS, during the treatment period. Opioid use will also be assessed using the Opioid 2000 ng tests on the UDS.
Time Frame: At week 6
Population: Intention to treat analysis was done including drop-out
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Stage 1 Placebo | Stage 1 AMC
Number analyzed (Participants) | 294 | 109
days
  Amphetamine | 41.89 (1.0) | 41.95 (0.3)
  Non-Methamphetamine Drug | 28.53 (14.7) | 31.47 (13.8)
  Cocaine | 41.87 (0.6) | 41.87 (0.5)
  Alcohol | 36.44 (9.5) | 37.89 (7.2)
  Cigarettes | 15.29 (18.7) | 16.31 (18.2)

15. Secondary Outcome: Mean Number of Abstinent Days of Participants Who Used Other Substance Measured by UDS at Stage 2
Description: as for outcome 14
Time Frame: at week 12
Population: As per study protocol, stage 2 secondary outcomes are reported for only re-randomized groups (Placebo and AMC)
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Stage 2 Re-Randomized Placebo | Stage 2 Re-Randomized AMC
Number analyzed (Participants) | 111 | 114
days
  Amphetamine | 44.96 (0.3) | 44.95 (0.3)
  Non-Methamphetamine drug | 30.99 (15.2) | 31.05 (16.1)
  Cocaine | 44.9 (0.4) | 44.88 (0.5)
  Alcohol | 38.41 (11.9) | 39.91 (9.1)
  Cigarettes | 17.11 (20.0) | 19.31 (20.1)

16. Secondary Outcome: Mean Change of Proportion of Other Substance Abstinent Days Measured by Self-report at Stage 1
Description: Proportion of abstinent days of other substance including Alcohol, Cigarettes and E- Cigarettes was measured by self-report on TLFB during the treatment period.
Time Frame: Baseline, week 6
Measure: Mean (Standard Error); unit: proportion of abstinent days
Arm/Group | Stage 1 Placebo | Stage 1 AMC
Number analyzed (Participants) | 294 | 109
proportion of abstinent days
  Alcohol | -0.054 (0.011) | -0.016 (0.017)
  Cigarettes | 0.054 (0.010) | 0.103 (0.021)
  E- Cigarettes | -0.064 (0.009) | -0.072 (0.016)

17. Secondary Outcome: Mean Change of Proportion of Other Substance Abstinent Days Measured by Self-report at Stage 2
Description: as for outcome 16
Time Frame: week 7, week 12
Population: as for outcome 11
Measure: Mean (Standard Error); unit: proportion of abstinent days
Arm/Group | Stage 2 Re-Randomized Placebo | Stage 2 Re-Randomized AMC
Number analyzed (Participants) | 111 | 114
proportion of abstinent days
  Alcohol | -0.035 (0.012) | -0.035 (0.016)
  Cigarettes | 0.038 (0.012) | 0.119 (0.022)
  E- Cigarettes | -0.057 (0.011) | -0.079 (0.014)

18. Secondary Outcome: Mean Change in Number of Other Substance Use by Self-report at Stage 1
Description: Number of other substance (Alcohol and Cigarettes) use was measured by self-report recall on Timeline Followback (TLFB) during the treatment period.
Time Frame: Baseline, week 6
Population: Intention to treat analysis was done including drop-out
Measure: Mean (Standard Error); unit: substances
Arm/Group | Stage 1 Placebo | Stage 1 AMC
Number analyzed (Participants) | 294 | 109
substances
  Alcohol | 0.358 (1.503) | -1.604 (3.290)
  Cigarettes | -12.642 (7.221) | -55.873 (14.154)

19. Secondary Outcome: Mean Change in Number of Other Substance Use by Self-report at Stage 2
Description: as for outcome 18
Time Frame: week 7, week 12
Population: As per study protocol, stage 2 secondary outcomes are reported for only re-randomized groups (Placebo and AMC). These numbers come from a model which does not use the Stage 2 Not rerandomized data so we do not have any estimates for the same.
Measure: Mean (Standard Error); unit: substances
Arm/Group | Stage 2 Re-Randomized Placebo | Stage 2 Re-Randomized AMC
Number analyzed (Participants) | 111 | 114
substances
  Alcohol | 1.695 (1.779) | -2.942 (3.121)
  Cigarettes | -9.925 (7.801) | -58.591 (14.594)

20. Secondary Outcome: Change in Proportion of E-cigarettes Abstinent Days by Self-report at Stage 1
Description: Proportion of abstinent days of E- Cigarettes was measured by self-report at stage 1.
Time Frame: Baseline, week 6
Measure: Mean (Standard Error); unit: Proportion of abstinent days
Arm/Group | Stage 1 Placebo | Stage 1 AMC
Number analyzed (Participants) | 294 | 109
Proportion of abstinent days | -0.064 (0.009) | -0.072 (0.016)

21. Secondary Outcome: Change in Proportion of E-cigarettes Abstinent Days by Self-report at Stage 2
Description: Proportion of abstinent days of E- Cigarettes was measured by self-report at stage 2.
Time Frame: week 7, week 12
Population: As per study protocol, stage 2 secondary outcomes are reported for only re-randomized groups (Placebo and AMC)
Measure: Mean (Standard Error); unit: Proportion of abstinent days
Arm/Group | Stage 2 Re-Randomized Placebo | Stage 2 Re-Randomized AMC
Number analyzed (Participants) | 111 | 109
Proportion of abstinent days | -0.057 (0.011) | -0.079 (0.014)

22. Secondary Outcome: Mean Change of Depression Symptom Score by PHQ-9 at Stage 1
Description: Patient Health Questionnaire-9 (PHQ-9) measures participants depression symptoms. Possible scores range from 0-27, with higher scores indicating a more severe depression symptoms.
  PHQ-9 scores reflect depression severity, ranges from 0-27 (0 no depressive symptoms, 1-4 minimal depression, 5-9 mild depression, 10-14 moderate depression, 15-19 moderately severe depression, 20-27 severe depression)
Time Frame: Baseline, week 6
Population: Intention to treat analysis was done including drop-out
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Stage 1 Placebo | Stage 1 AMC
Number analyzed (Participants) | 294 | 109
score on a scale | -3.26 (0.34) | -4.78 (0.70)

23. Secondary Outcome: Mean Change of Depression Symptom Score by PHQ-9 at Stage 2
Description: Patient Health Questionnaire-9 measures participants depression symptoms. Possible scores range from 0-27, with higher scores indicating a more severe depression symptoms.
  PHQ-9 scores reflect depression severity, ranges from 0-27 (0 no depressive symptoms, 1-4 minimal depression, 5-9 mild depression, 10-14 moderate depression, 15-19 moderately severe depression, 20-27 severe depression)
Time Frame: week 7, week 12
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stage 2 Re-Randomized Placebo | Stage 2 Re-Randomized AMC
Number analyzed (Participants) | 111 | 114
score on a scale | -3.66 (0.37) | -4.39 (0.64)

24. Secondary Outcome: Mean Change of Quality of Life (QOL) by PhenX Core Tier 1 Instrument at Stage 1
Description: Mean change score of QOL (General health, Physical health, and Mental health) from baseline will be assessed by PhenX (Phenotypes and eXposures) Core Tier 1 instrument: Quality of Life (QOL), which measures participants' quality of life during the past 30 days. Possible scores range from 0 to 30 (number of days in the past 30 in which health was good), with higher scores indicating a better quality of life.
Time Frame: Baseline, Week 6
Population: Intention to treat analysis was done including drop-out
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Stage 1 Placebo | Stage 1 AMC
Number analyzed (Participants) | 294 | 109
score on a scale
  Physical Health | 1.013 (0.805) | 1.425 (1.225)
  Mental Health | 1.071 (0.842) | 3.785 (1.380)
  General Health | -1.168 (0.957) | 1.582 (1.442)

25. Secondary Outcome: Mean Change of Quality of Life (QOL) by PhenX Core Tier 1 Instrument at Stage 2
Description: Mean change score of QOL (General health, Physical health, and Mental health) from baseline will be assessed by PhenX Core Tier 1 instrument: Quality of Life (QOL), which measures participants' quality of life during the past 30 days. Possible scores range from 0 to 30 (number of days in the past 30 in which health was good), with higher scores indicating a better quality of life.
Time Frame: week 7, week 12
Population: As per study protocol, stage 2 secondary outcomes are reported for only re-randomized groups (Placebo and AMC)
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Stage 2 Re-Randomized Placebo | Stage 2 Re-Randomized AMC
Number analyzed (Participants) | 111 | 114
score on a scale
  Physical Health | 0.877 (0.870) | 1.561 (1.147)
  Mental Health | 2.035 (0.917) | 2.821 (1.345)
  General Health | 0.262 (1.038) | 0.152 (1.365)

26. Secondary Outcome: Mean Change of Overall Functioning as Measured by Treatment Effectiveness Assessment (TEA) at Stage 1
Description: The Treatment Effectiveness Assessment is a 4-item self-administered assessment that uses a Likert scale (1-10) to document changes in four life domains: substance use, health, lifestyle, and community and is collected at screening, mid-treatment (Week 6 Visit 2) and end-of-treatment (Week 12 Visit 2).
  Possible scores range from 4-40, with higher scores indicating a higher overall functioning.
Time Frame: Baseline, week 6
Population: Intention to treat analysis was done including drop-out
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Stage 1 Placebo | Stage 1 AMC
Number analyzed (Participants) | 294 | 109
score on a scale | 2.2 (1.0) | 6.5 (1.5)

27. Secondary Outcome: Mean Change of Overall Functioning as Measured by Treatment Effectiveness Assessment (TEA) at Stage 2
Description: as for outcome 26
Time Frame: week 7, week 12
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stage 2 Re-Randomized Placebo | Stage 2 Re-Randomized AMC
Number analyzed (Participants) | 111 | 114
score on a scale | 2.5 (1.1) | 6.2 (1.5)

28. Secondary Outcome: Number of Participants Who Completed the Visit in Week 12
Time Frame: At week 12
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 2 Re-Randomized Placebo | Stage 2 Re-Randomized AMC | Stage 2 Not Re-Randomized Placebo | Stage 2 Not Re-Randomized AMC
Number analyzed (Participants) | 111 | 114 | 69 | 109
Participants | 106 | 103 | 28 | 78

29. Secondary Outcome: Participant Satisfaction Rating Measured by Study Satisfaction Survey at the End of the Study
Description: The Study satisfaction survey measures participants satisfaction. We do not have a proper score range (varied range with some free text questions also)
Time Frame: At week 12
Population: We did not collect data about satisfaction.
Arm/Group | Stage 1 Placebo | Stage 1 AMC | Stage 2 Re-Randomized Placebo | Stage 2 Re-Randomized AMC | Stage 2 Not Re-Randomized Placebo | Stage 2 Not Re-Randomized AMC
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline to 12 weeks
Arm/Group | Stage 1 Placebo | Stage 1 AMC | Stage 2 Re-Randomized Placebo | Stage 2 Re-Randomized AMC | Stage 2 Not Re-Randomized Placebo | Stage 2 Not Re-Randomized AMC
All-Cause Mortality (participants affected / at risk) | 0/294 | 0/109 | 0/111 | 0/114 | 0/69 | 0/109
Serious Adverse Events (participants affected / at risk) | 4/294 | 1/109 | 4/111 | 3/114 | 1/69 | 3/109
Other Adverse Events (participants affected / at risk) | 45/294 | 41/109 | 8/111 | 32/114 | 0/69 | 6/109
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stage 1 Placebo (N=294) | Stage 1 AMC (N=109) | Stage 2 Re-Randomized Placebo (N=111) | Stage 2 Re-Randomized AMC (N=114) | Stage 2 Not Re-Randomized Placebo (N=69) | Stage 2 Not Re-Randomized AMC (N=109)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Substance-induced psychotic disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paranoia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Victim of crime (Social circumstances) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Stage 1 Placebo (N=294) | Stage 1 AMC (N=109) | Stage 2 Re-Randomized Placebo (N=111) | Stage 2 Re-Randomized AMC (N=114) | Stage 2 Not Re-Randomized Placebo (N=69) | Stage 2 Not Re-Randomized AMC (N=109)
Nausea (Gastrointestinal disorders) | 45 | 41 | 8 | 32 | 0 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2019-01-31): https://cdn.clinicaltrials.gov/large-docs/75/NCT03078075/Prot_000.pdf
  • Statistical Analysis Plan (2019-09-13): https://cdn.clinicaltrials.gov/large-docs/75/NCT03078075/SAP_001.pdf
  • Informed Consent Form (2018-12-19): https://cdn.clinicaltrials.gov/large-docs/75/NCT03078075/ICF_002.pdf